CLINICAL TRIAL: NCT06619808
Title: Efficacy and Safety of Hyperbaric Oxygen Therapy in Adult Metabolic Dysfunction-associated Steatotic Liver Diseases (MASLD) Patients : a Randomized Controlled Trial
Brief Title: Hyperbaric Oxygen Therapy for Metabolic Dysfunction-associated Steatotic Liver Diseases
Acronym: MASLD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jinling Hospital, China (Other)
Responsible Party: Principal Investigator, Lu Chen, MS, Jinling Hospital, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024DZKY-052-01
Record Dates: First submitted 2024-08-11; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Metabolic Dysfunction-associated Steatotic Liver Disease; Hepatic Steatosis; Non-alcoholic Fatty Liver Diseases
Keywords: Metabolic Dysfunction-associated Steatotic Liver Disease; Hyperbaric Oxygen Therapy; Non-alcoholic Fatty Liver Diseases; Oxygen Therapy
MeSH Terms: conditions — Fatty Liver | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hyperbaric Oxygen Therapy (Experimental): Participants receive 20 session of hyperbaric oxygen therapy (HBOT) in 1 month (inhalation of 100% oxygen in a pressure chamber under 2.0 ATA for 60 minutes).
  Interventions: Procedure: Hyperbaric oxygen therapy
- Symptomatic Treatment (No Intervention): Participants receive basic symptomatic treatments like antidiabetic drug, antihypertensive drug, and hepatic protector.

INTERVENTIONS:
Procedure: Hyperbaric oxygen therapy — Participants receive 20 session of hyperbaric oxygen therapy (HBOT) in one month (inhalation of 100% oxygen in a pressure chamber under 2.0 ATA for 60 minutes).
  Arms: Hyperbaric Oxygen Therapy

SUMMARY:
The goal of this clinical trial is to learn if hyperbaric oxygen therapy (HBOT) works to treat Metabolic Dysfunction-associated Steatotic Liver Diseases (MASLD). The main questions it aims to answer are:

Does HBOT decreases the fat content and fibrosis state of liver in adult MASLD patients? Does HBOT improves the liver function and metabolic condition in adult MASLD patients?

Participants will:

Receive HBOT for 20 times in 1 month or recerive regular drug; Visit the clinic for checkups and tests at the starting, ending of the therapy and 6 month after the therapy.

DETAILED DESCRIPTION:
Metabolic Dysfunction-associated Steatotic Liver Diseases (MASLD) patients who meet our principles would be randomized into 2 groups: the HBOT group and CON group. The entire project is not blinded. In HBOT group, participants will receive HBOT for 20 times in 1 month (2.0ATA, 60min), which is the common setting in clinical use.The CON group, which means the control group, recerives regular drug, like liver-protective drugs and hypoglycemic drugs. The visiting times are week 0 (starting of the project), week 4 (ending of the therapy), week 28 (6 months after the therapy), when participants get checkups and tests. The primary outcome of our study are the change of liver fat content and stiffness in Fibroscan. The secondary outcomes invovle changes of liver function enzymes and metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Metabolic dysfunction-associated steatotic liver disease patients

Exclusion Criteria:

* Participants are unfit for hyperbaric treatment.
* Participants with prior oxygen therapy within the last 6 months.
* Participants with history of viral hepatitis, hemochromatosis, Wilson disease, autoimmune hepatitis, primary biliary cirrhosis, sclerosing cholangitis, biliary obstruction, alpha-1 antitrypsin deficiency.
* Participants with severe organ dysfunctions or malignant tumors.
* Participants have weight loss plan or major operations within the last 6 months.
* Participants are unable to provide informed consent or currently participating in or has within the last 3 months participated in any other clinical trial.
* Participants are pregnant or lactating.
* Participants with claustrophobia or that cannot decompress properly.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-07-29 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Change of liver stiffness | Before the 1-month treatment, directly after the treatment, 6 months after the treatment
  We use E value to describe liver stiffness by Fibroscan noninvasive transient elastography.
Change of liver fat content | Before the 1-month treatment, directly after the treatment, 6 months after the treatment
  We use controlled attenuation parameter (CAP) to evaluate liver fat content by Fibroscan noninvasive transient elastography.

SECONDARY OUTCOMES:
Change of liver enzymes | Before the 1-month treatment, directly after the treatment, 6 months after the treatment
  Alanine aminotransferase (ALT), aspertate aminotransferase(AST)
Change of fasting blood glugose | Before the 1-month treatment, directly after the treatment, 6 months after the treatment
Change of fasting insulin | Before the 1-month treatment, directly after the treatment, 6 months after the treatment
Change of cholesterol | Before the 1-month treatment, directly after the treatment, 6 months after the treatment
  total cholesterol (TC), low density lipoprotein (LDL-C), high density lipoprotein(HDL-C)
change of total triglyceride | Before the 1-month treatment, directly after the treatment, 6 months after the treatment
  TG

OTHER OUTCOMES:
Safety of hyperbaric oxygen therapy | After each session of HBOT and up to 6 months after the HBOT therapy.
  We conduct questionnaires of adverse reaction after every therapy time and follow-up visit.

CONTACTS AND LOCATIONS:
Overall Officials: Miaofang Yang, MD, Study Director — General Hospital of Eastern Theater Command, China
Locations (1):
- General Hospital of Eastern Theater Command, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
Not suitable